CLINICAL TRIAL: NCT04948242
Title: Epidemiologic, Clinical Characteristics and Risk Factors of Critical Ill Patients Admitted to the ICU for Severe Acute Respiratory Syndrome Coronavirus 2 Infection (COVID-19)
Brief Title: Characteristics of Critically Ill Patients With Severe Acute Respiratory Syndrome Coronavirus 2 Infection (COVID-19)
Acronym: GETCOV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Collaborators: Sociedad Española de Medicina Intensiva,critica y unidades coronarias (Unknown)
Responsible Party: Principal Investigator, Alejandro Rodriguez Oviedo , MD, MD,PhD,MsC, Hospital Universitari Joan XXIII de Tarragona.
Other Study IDs: COVID-19/SEMICYUC
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV2 Infection
Keywords: COVID-19; Severe SARS-CoV-2 infection; Critically ill patients; ADRS; Viral pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive critically ill patients admitted to ICU with severe SARS-CoV-2 infection: Consecutive adult patients (> 16 years) with laboratory confirmed SARS-CoV-2 infection, detected by RT-PCR positive test of nasopharyngeal, oropharyngeal , swab or invasive respiratory samples according to the WHO recommendations. The follow-up of patients was to ICU discharge or death whichever occurred first. No interventions will be made. Only anonymized demographic data, clinical data, laboratory data and ventilatory support data will be collected. There is no standardized pharmacological treatment protocol. Only basic data are collected about the different treatments administered by the attending physician.

SUMMARY:
A multicenter observational, prospective cohort study that consisted of a large-scale data source of hospital ICU admissions and patient-level clinical data in Spain.

The main objective is to develop a national database belonging to SEMICYUC (Spanish Society of Critical Care) to describe epidemiological and clinical characteristics and risk factors related to ICU mortality in critically ill patients admitted to ICU due to severe COVID-19 in Spain.

DETAILED DESCRIPTION:
Design: A multicenter observational, prospective cohort study

Setting: Intensive Care Units

Subjects: Adult Critical patients admitted to ICU with severe community-acquired pneumonia due to confirmed SARS CoV-2 infection (COVID-19).

Data Collection and Validation Data was obtained from a voluntary registry created by Spanish Society of Intensive Care Medicine-SEMICYUC. All consecutive cases admitted to the ICU were collected.

There were no patients excluded from the analysis that was enrolled to participating ICU and met criteria.

Data were collected using a paper CRF (case Report Form). CRF collect and record all protocol-required information, which is transcribed from patient source documents, such as hospital records and laboratory reports during the patient's participation in the study. Before being sent to the National Study Coordinator (AR) this data was de-identified (not traceable to the patient) by removing the patient's name, medical record number, etc., and giving the patient a unique study number. We implemented a double data entry model for potential errors in real-time. Data was entered twice by two different Data Entry personnel based on the same set of data collected in the paper CRFs. All data were reviewed, and values that appeared incongruent or out of range were manually validated by confirming the accuracy of the data with the Study Coordinator (AR). The database was validated and cleaned before the statistical analysis and the study database was locked to prevent any further changes, and to ensure data consistency and integrity for the statistical reporting and analysis.

Sample size calculation:

No statistical sample size calculation was performed a priori, and sample size was equal to the number of patients admitted to the participant's ICUs with confirmed COVID-19 during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Severe community-acquired pneumonia due SARS CoV-2 infection and acute respiratory failure with microbiological confirmation (RT-PCR) according international guidelines
2. Age >= 16 years without upper limit

Exclusion Criteria:

1. Age < 16 years
2. Patients with SARS-CoV-2 infection without acute respiratory failure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients with community-acquired pneumonia due to SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic and Clinical Characteristics and risk factors for ICU mortality in critically ill patients with COVID-19 in Spain | Observational period from ICU admission to data of discharge alive or date of death from any cause at days 28 of ICU length of stay and ICU discharge
  To determine demographics and clinical factors associated with ICU mortality at days-28 and ICU discharge

SECONDARY OUTCOMES:
Support respiratory type and prognosis | Observational period from ICU admission to data of discharge alive or date of death from any cause at days 28 of ICU length of stay and ICU discharge
  Association between respiratory support used at ICU admission and ICU mortality
Comorbidities and prognosis | Observational period from ICU admission to data of discharge alive or date of death from any cause at days 28 of ICU length of stay and ICU discharge
  Association between different comorbidities (diabetes, obesity, hypertension, etc) and ICU mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rodriguez Oviedo, MD,PhD,MsC, Study Director — Hospital Universitari de Tarragona Joan XXIII
Locations (1):
- Hospital Universitario de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berenguer J, Ryan P, Rodriguez-Bano J, Jarrin I, Carratala J, Pachon J, Yllescas M, Arriba JR; COVID-19@Spain Study Group; Fundacion SEIMC-GESIDA; Hospital General Universitario Gregorio Maranon; Hospital Universitario La Paz; Hospital Infanta Leonor; Complejo Hospitalario Virgen de la Salud; Hospital Universitario Rafael Mendez; Hospital Universitario de Cruces; Hospital de Melilla; Hospital San Eloy de Barakaldo; Hospital Universitario Central de Asturias; Hospital General Universitario de Alicante; Hospital Virgen de la Victoria; Hospital Universitario Puerto Real; EOXI Pontevedra e Salnes; Hospital de Figueres; Hospital Sant Jaume de Calella; Hospital del Mar; Hospital Virgen de la Arrixaca; Hospital de Can Misses; Hospital de Sagunto; Hospital Clinico San Cecilio; Hospital Universitario Principe de Asturias; Parc Sanitari Sant Joan de Deu; Hospital Nuestra Senora de Gracia; HC Marbella Internacional Hospital; Hospital La Princesa; Hospital Josep Trueta; Hospital Dos de Maig; Hospital Arnau de Vilanova-Lliria; Hospital General Universitario de Elche; Hospital Clinico Universitario de Valencia; Complejo Asistencial de Avila; Hospital Comarcal de Alcaniz; Hospital Universitario Marques de Valdecilla; Hospital Quiron-Salud de Torrevieja; Hospital Universitario Miguel Servet; SCIAS, Hospital de Barcelona; Fundacion Hospital Universitario Alcorcon; Hospital Alvaro Cunqueiro; Complejo Asistencial Universitario de Salamanca; Hospital Universitario Severo Ochoa; Hospital CIMA-Sanitas; Hospital HLA Inmaculada; Hospital Universitario Rio Hortega; Hospital de Guadalajara; Hospital Universitario Infanta Sofia; Hospital Comarcal de Blanes; Hospital Universitari de Tarragona Joan XXIII; Hospital Universitario Basurto; Hospital Universitario de Canarias; Hospital Universitario de Gran Canaria Dr Negrin; Hospital Son Espases; Hospital Universitario de Mostoles; Complejo Hospitalario Universitario A Coruna; Hospital Costa del Sol; Hospital Clinico Universitario Lozano Blesa; Hospital Mutua de Terrassa; Hospital de la Plana; Hospital Virgen de la Concha-Complejo Asistencial de Zamora; Complejo Hospitalario Universitario Insular Materno-Infantil; Hospital de la Marina Baixa; Hospital Universitario Virgen Macarena; Hospital Universitari de Bellvitge; Hospital Universitario y Politecnico la Fe; Hospital Universitario del Vinalopo; Hospital de Sabadell (Parc Tauli); Hospital Clinic de Barcelona; Hospital Universitario de la Ribera; Fundacion Jimenez Diaz; Hospital Clinico Universitario de Valladolid; Hospital Clinico San Carlos; Hospital Santa Creu i Sant Pau; Clinica Universitaria de Navarra-Campus Madrid; Hospital Son Llatzer; Hospital General de la Defensa Gomez Ulla; Hospital Universitario de Alava; Hospital Santos Reyes; Hospital Dr Jose Molina Orosa; Hospital Vall d'Hebron; Hospital Universitario Rey Juan Carlos; Complejo Hospitalario Universitario Santa Lucia; Hospital Santa Barbara; Complejo Hospitalario Universitario de Ferrol; Hospital de l'Esperit Sant; Hospital Universitario los Arcos del Mar Menor; Hospital HLA Universitario Moncloa; Hospital Virgen del Puerto; Hospital Marina Salud de Denia; Hospital Universitario de Jerez; Hospital Reina Sofia de Tudela; Hospital Clinico Universitario de Santiago de Compostela; Hospital Universitario del Henares; Hospital Universitario Lucus Augusti; Hospital de Donostia; Hospital de Urduliz Alfredo Espinosa; Hospital de Mendaro; Hospital Juan Ramon Jimenez; Hospital de Tortosa Virgen de la Cinta; Hospital Riotinto; Hospital Vega Baja; Hospital Puerta de Hierro; Hospital Universitario de Getafe; Hospital General de la Palma; Hospital El Bierzo; Fundacion Hospital de Calahorra; Hospital Alto Deba; Hospital Universitario San Juan de Alicante; Hospital de Guadarrama; Hospital Universitario de Jaen; Hospital de Mataro; Hospital de Palamos; Hospital Universitario de Valme; Clinica Universitaria de Navarra-Campus Navarra; Hospital Clinica Benidorm; Hospital Doce de Octubre; Hospital Universitario Virgen del Rocio; Hospital Universitario Ramon y Cajal; Hospital Universitario San Pedro; Hospital Quiron A Coruna; HM Sanchinarro; Hospital Francesc de Borja; Complejo Hospitalario Universitario Nuestra Senora de La Candelaria; Hospital Universitario HM Monteprincipe; Hospital Universitario HM Puerta del Sur; Hospital Universitario HM Torrelodones; Hospital Universitario HM Madrid; Hospital Don Benito-Villanueva de la Serena; Hospital de Viladecans; Centro Nacional de Epidemiologia. Characteristics and predictors of death among 4035 consecutively hospitalized patients with COVID-19 in Spain. Clin Microbiol Infect. 2020 Nov;26(11):1525-1536. doi: 10.1016/j.cmi.2020.07.024. Epub 2020 Aug 4. PMID 32758659
- [Background] Berenguer J, Borobia AM, Ryan P, Rodriguez-Bano J, Bellon JM, Jarrin I, Carratala J, Pachon J, Carcas AJ, Yllescas M, Arribas JR; COVID-19@Spain and COVID@HULP Study Groups. Development and validation of a prediction model for 30-day mortality in hospitalised patients with COVID-19: the COVID-19 SEIMC score. Thorax. 2021 Sep;76(9):920-929. doi: 10.1136/thoraxjnl-2020-216001. Epub 2021 Feb 25. PMID 33632764
- [Result] Rodriguez A, Ruiz-Botella M, Martin-Loeches I, Jimenez Herrera M, Sole-Violan J, Gomez J, Bodi M, Trefler S, Papiol E, Diaz E, Suberviola B, Vallverdu M, Mayor-Vazquez E, Albaya Moreno A, Canabal Berlanga A, Sanchez M, Del Valle Ortiz M, Ballesteros JC, Martin Iglesias L, Marin-Corral J, Lopez Ramos E, Hidalgo Valverde V, Vidaur Tello LV, Sancho Chinesta S, Gonzales de Molina FJ, Herrero Garcia S, Sena Perez CC, Pozo Laderas JC, Rodriguez Garcia R, Estella A, Ferrer R; COVID-19 SEMICYUC Working Group. Deploying unsupervised clustering analysis to derive clinical phenotypes and risk factors associated with mortality risk in 2022 critically ill patients with COVID-19 in Spain. Crit Care. 2021 Feb 15;25(1):63. doi: 10.1186/s13054-021-03487-8. PMID 33588914
- [Derived] Manrique S, Claverias L, Magret M, Masclans JR, Bodi M, Trefler S, Canadell L, Diaz E, Sole-Violan J, Bisbal-Andres E, Natera RG, Moreno AA, Vallverdu M, Ballesteros JC, Socias L, Vidal FG, Sancho S, Martin-Loeches I, Rodriguez A. Timing of intubation and ICU mortality in COVID-19 patients: a retrospective analysis of 4198 critically ill patients during the first and second waves. BMC Anesthesiol. 2023 Apr 27;23(1):140. doi: 10.1186/s12871-023-02081-5. PMID 37106321
- See also: Spanisho Society of Critical Care web — https://semicyuc.org/covid-19/